CLINICAL TRIAL: NCT01565837
Title: Phase II Evaluation of Concurrent Ipilimumab Therapy and Stereotactic Ablative Radiation Therapy (SART) for Oligometastatic But Unresectable Malignant Melanoma
Brief Title: Concurrent Ipilimumab and Stereotactic Ablative Radiation Therapy (SART) for Oligometastatic But Unresectable Melanoma
Acronym: SART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfram Samlowski (Other)
Collaborators: Comprehensive Cancer Centers of Nevada (Other)
Responsible Party: Sponsor-Investigator, Wolfram Samlowski, Physician, Comprehensive Cancer Centers of Nevada; Member, Developmental Therapeutics and Genitourinary Committee, US Oncology Research; Clinical Professor, University of Nevada, Reno, Comprehensive Cancer Centers of Nevada
Organization: Comprehensive Cancer Centers of Nevada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMS CA184-168
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Melanoma
Keywords: Melanoma; Malignant Melanoma; Metastatic; Oligometastatic; Radiosurgery; Radiosurgery, Stereotactic; Stereotactic Radiosurgery; Ipilimumab; Yervoy; MDX-010; Circulating Tumor Cells
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Neoplastic Cells, Circulating | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab + SART (Experimental): Patients with oligometastatic but unresectable malignant melanoma will receive induction ipilimumab plus concurrent SART followed by maintenance ipilimumab.
  Interventions: Drug: Ipilimumab; Radiation: Stereotactic Ablative Radiosurgery (SART)

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 10mg/kg administered intravenously over 90-minute period every 3 weeks for a total of four doses as tolerated. Maintenance ipilimumab (10 mg/kg intravenously every 3 months) will be administered beginning Week 24, as long as there is clinical benefit in the opinion of the investigator using immune related response criteria, and there are no novel or unexpected Grade 3 or 4 toxicities.
  Other Names: Yervoy; MDX-010
Radiation: Stereotactic Ablative Radiosurgery (SART) — Definitive radiotherapy will be administered to up to 1-5 lesions using SART techniques after initial dose of ipilimumab. Radiotherapy will be timed before start of 3rd cycle of ipilimumab treatment to maximize synergy (week 6).

SUMMARY:
The purpose of this study is to evaluate if precisely-targeted radiation therapy, known as stereotactic ablative radiotherapy (SART), given during treatment with the drug ipilimumab (Yervoy) will improve survival for patients with melanoma that has spread to five or fewer sites (oligometastatic).

Blood samples will be collected for research purposes. Planned studies include exploration of certain gene mutations and serum markers as predictors of response to ipilimumab treatment. Research lab studies will also evaluate if circulating tumor cells (CTC) can be accurately detected and isolated from the blood using novel laboratory techniques and if they are a prognostic/predictive marker for treatment response. Test results will not be given to participants or their physicians. In some cases, CTC may be grown for long-term cell lines for further research.

DETAILED DESCRIPTION:
Primary Objectives:

1. To evaluate the effectiveness of concurrent ipilimumab therapy and SART of melanoma based on 1-year and 2-year overall survival.
2. To evaluate the safety and tolerability of concurrent ipilimumab therapy and SART of melanoma based on CTCAE grading of toxicities, and to identify any novel or unexpected Grade 3 or 4 toxicities thought specifically related to ipilimumab and concurrent SART during first 3 cycles of ipilimumab therapy (prior to week 9) in a Phase II study.

Secondary Objectives:

1. To evaluate the 1-year and 2-year disease control rates (CR+PR+SD)
2. Assess treatment response based on Immune Related Response Criteria (irRC) and mWHO criteria.
3. Characterize overall survival by Kaplan-Meier analysis.

Exploratory Objectives:

1. Evaluate individual lesion control (<25% progression) following body SART at 6, 12, 24 months.
2. Describe number of patients requiring retreatment of any local lesion with surgery or other treatments.
3. Describe the incidence of new brain metastases following ipilimumab therapy.
4. Describe the incidence of treatment related toxicity and/or symptomatic bleeding, perforation, or necrosis at SART treated tumor sites.
5. Explore the use of circulating melanoma cells and serum metastasis gene expression levels as prognostic and predictive (intermediate) markers to identify responding patients.
6. Assess the effect of therapy on quality of life, using ECOG score as a surrogate.

Study Rationale:

Ipilimumab may markedly enhance the immunologic responses to tumor antigen released from necrotic tumor cells by radiotherapy by promoting cytotoxic T cell activation, while preventing induction of antigen tolerance. In addition, further beneficial immunologic effects may be achieved by the reduction in the amount of viable tumor cell mass. The net effect may be to promote a significantly enhanced antitumor T cell response. This will result in improved 1-year and 2-year survival, especially if a minimal or microscopic disease state can be achieved within a patient following SART.

Biologic Correlation Studies:

There are currently no standard prognostic or predictive markers to evaluate or predict outcome of ipilimumab therapy. This study provides the opportunity for exploratory analysis of several candidate hypotheses that may predict outcome.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV melanoma (AJCC 6th edition) with 5 or less metastatic sites that are not amenable to curative surgical resection, but can be adequately delineated for SART
* All sites of metastatic disease acceptable except brain-only and eye metastases, provided SART can be safely delivered to the site.
* Up to 2 prior systemic treatments for metastatic disease.
* Mucosal or ocular melanoma is allowed.
* Radiotherapy consultation and insurance preapproval for SART prior to enrollment.
* CT or MRI within 28 days of enrollment showing no evidence of brain metastases. Brain metastases allowed if stable by scans for ≥ 28 days following treatment.
* CT, PET/CT or MRI scan of chest, abdomen, pelvis (and soft tissue as indicated); bone scan (as indicated); and photographs of skin lesions (if applicable) within 28 days of enrollment.
* Hematology, liver function and renal function lab tests within required parameters.
* Recovered from all prior surgery and/or adjuvant treatment.
* No active or chronic infection with HIV, Hepatitis B or Hepatitis C.
* ECOG Performance Status 0 or 1.
* Men and women ≥ 18 years old.
* Men/Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

* Untreated or uncontrolled brain metastases.
* Prior treatment with CTLA-4 agent, PD-1 or PD-1 ligand mAb or inhibitor for metastatic disease or as adjuvant therapy (or participation in blinded study).
* History of melanoma-associated retinopathy.
* History of other active malignancy within last 2 years, except adequately treated basal cell carcinoma or squamous cell skin cancer or carcinoma in situ of cervix, unless disease-free for 2 years.
* Autoimmune disease (vitiligo is not a basis for exclusion).
* History of clinically active diverticulitis (diverticulosis is not exclusion criterion per se).
* Serious uncontrolled medical disorder or active infection that would impede treatment.
* Underlying medical or psychiatric condition that would cause administration of ipilimumab to be hazardous, or would obscure interpretation of AEs.
* Any non-oncology vaccine therapy up to 1 month before or after any dose of ipilimumab.
* Concomitant therapy with IL-2, interferon, other non-study immunotherapy, or cytotoxic chemotherapy; immune-suppressive agents within 30 days of registration; other investigational therapies; chronic use of systemic corticosteroids (however, a low stable dose steroid for mild brain edema or adrenal insufficiency is allowed; topical and inhaled standard dose corticosteroids are allowed).
* Dementia or significantly altered mental status that would prohibit understanding or rendering of informed consent and compliance with protocol requirements.
* Pregnant or breastfeeding women.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g. infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of concurrent ipilimumab and SART - Acute Toxicity | Week 9
Safety and tolerability of concurrent ipilimumab and SART - Subacute Toxicity | Week 15

SECONDARY OUTCOMES:
1-year disease control rates (CR+PR+SD) based on irRC and mWHO criteria | 2 year minimum follow up on study participants
2-year disease control rates (CR+PR+SD) based on irRC and mWHO criteria | 2 year minimum follow up on study participants
1-year overall survival | 2 year minimum follow up on study participants
2-year overall survival | 2 year minimum follow up on study participants

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Samlowski, MD, Principal Investigator — Comprehensive Cancer Centers of Nevada
Locations (1):
- Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada, United States